CLINICAL TRIAL: NCT03880981
Title: NSAID Use and Healing After Tibia Fractures and Achilles Tendon Ruptures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Vanessa Franco, MD, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VFranco
Record Dates: First submitted 2019-02-22; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Musculoskeletal Injury
Keywords: fracture; tendon rupture; NSAID; healing
MeSH Terms: conditions — Fractures, Bone | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Active Comparator): Patients will receive 650mg PO Acetaminophen every 6 hours as needed for pain
  Interventions: Drug: Acetaminophen
- Ibuprofen (Active Comparator): Patients will receive 600mg PO Ibuprofen every 6 hours as needed for pain
  Interventions: Drug: Ibuprofen 600 mg

INTERVENTIONS:
Drug: Ibuprofen 600 mg — ibuprofen 600mg Po q 6 hours prn pain
  Arms: Ibuprofen
Drug: Acetaminophen — acetaminophen 600mg po q6 hours prn pain
  Arms: Acetaminophen

SUMMARY:
Rationale: The Emergency Department (ED) typically serves as the front line for patients with acute fractures and tendon ruptures. Pain control for these patients is an essential task of the ED physician. With the advent of the opioid epidemic, ED physicians are becoming more inclined to prescribe non-narcotic pain medications such as non-steroidal anti-inflammatory drugs (NSAIDs). Yet, the effects of NSAIDs on musculoskeletal healing are controversial. The few human studies examining the effects of NSAID use on fracture healing have provided conflicting results. Even less is known about the effects of NSAIDs on tendon healing as this information has largely been gleaned from rodent studies with contradictory findings. There has never been a large, prospective, randomized, double-blinded study to determine the effects of NSAIDs on healing after fractures or tendon ruptures. Here, I propose to pilot the first prospective, randomized, double-blinded study examining the effects of NSAID use on healing after tibia fractures and Achilles tendon ruptures.

Aim 1 seeks to determine whether NSAID use is associated with an increased incidence of fracture nonunion and worse functional recovery six months following tibia fractures. I hypothesize that NSAID use after tibia fractures will be associated with an increased incidence of fracture nonunion and worse functional recovery. Aim 2 seeks to determine whether NSAID use is associated with worse functional recovery six months after Achilles tendon ruptures. I hypothesize that NSAID use after Achilles tendon ruptures will be associated with worse functional recovery.

Significance: Emergency Department providers commonly prescribe NSAIDs for pain control following fractures and tendon injuries. However, the implications of this practice on bone and tendon healing are unknown. This proposal will pilot the first prospective, randomized, double-blinded study to determine whether NSAID use affects healing after tibia fractures and Achilles tendon ruptures. Results from this study will impact NSAID prescribing patterns for tibia fractures and Achilles tendon ruptures in the ED, either by demonstrating that they impair recovery and should be avoided, or that they need not be withheld as an effective non-narcotic form of pain control.

DETAILED DESCRIPTION:
Specific Aims The Emergency Department (ED) typically serves as the front line for patients with fractures and tendon ruptures. Pain control for these patients is an essential task of the ED physician. With the advent of the opioid epidemic, ED physicians are becoming more inclined to prescribe non-narcotic pain medications such as non-steroidal anti-inflammatory drugs (NSAIDs). Yet, the effects of NSAIDs on musculoskeletal healing are highly controversial. There is some evidence that NSAIDs may prevent osteoblasts from rebuilding bone after fractures by inhibiting COX-2. Indeed, some retrospective studies have found NSAID use to be associated with an increased incidence of fracture nonunion after acetabular, tibial, and humeral shaft fractures, while other studies reported no difference. The only prospective randomized controlled trials evaluating the effects of NSAIDs on fracture healing reported no effect of NSAID use on healing after Colles fractures; however, these trials were likely underpowered to detect a difference in nonunion rates. Here, I propose to pilot the first large, prospective, randomized, double-blinded study examining the effects of NSAIDs on healing after tibia fractures, which are vulnerable to nonunion.

Similar to fractures, the effects of NSAIDs on tendon healing are unclear. Some studies suggest that NSAIDs may inhibit proliferation and migration of tendon cells after injury, while other studies indicate that NSAIDs enhance collagen synthesis. Rodent studies are equally conflicting, with some reports of worse outcomes associated with NSAID use and other studies showing no difference. Recently, I obtained preliminary data showing that NSAID use after Achilles tendon ruptures is associated with worse functional outcomes as measured by the Achilles Tendon Total Rupture Score (ATRS). While this was the first study examining the effects of NSAID use on recovery after Achilles tendon rupture in humans, the data were retrospective, observational, and not blinded. Here, I propose to pilot the first prospective, randomized, double-blinded study to determine the effects of NSAIDs on recovery after Achilles tendon ruptures.

Aim 1: Determine whether NSAID use is associated with an increased incidence of fracture nonunion and worse functional recovery six months after tibia fractures.

Hypothesis: I hypothesize that NSAID use after tibia fractures will be associated with an increased incidence of fracture nonunion and worse functional recovery.

Aim 2: Determine whether NSAID use is associated with worse functional recovery six months after Achilles tendon ruptures.

Hypothesis: I hypothesize that NSAID use after Achilles tendon ruptures will be associated with worse functional recovery.

Experimental Approach: Adult patients (18 years old and over) presenting to either the University of California Los Angeles (UCLA) Ronald Regan Emergency Department, the UCLA Santa Monica Emergency Department, or the UCLA Orthopedic after hours acute care clinic within 24 hours of sustaining a tibia fracture or Achilles tendon rupture will be screened for eligibility to participate. Patients will be excluded if they have a contraindication to Ibuprofen or Acetaminophen use, if they do not have access to e-mail, if they do not wish to participate, if they require emergent surgery (such as an open fracture), if they have a diagnosis of osteoporosis, or if they have already taken pain medication since their injury. Pregnant women will be excluded due to their inability to take NSAIDs. Children will be excluded due to differences in bone and tendon healing. The ED represents the optimal environment in which to conduct this study because most patients will initially present acutely to the ED with these injuries, often before taking any pain medication.

If patients elect to participate, they will be randomized to receive either Ibuprofen (600mg by mouth every 6 hours as needed for pain) or Acetaminophen (650 mg by mouth every 6 hours as needed for pain). I will use a permuted block design to develop the randomization schedule. Randomization will be stratified by sex. Sealed envelopes will be used to conceal the allocation. The treating physician will open the envelope and provide the assigned study medication and prescription bottle at discharge. Patients will be provided a one-month supply of their assigned pain medication. Patients and providers will be blinded to which medication the patient received. The individual medication capsules will be formulated to lack identifying information. Study coordinators will record the patients' randomly generated study identification number and prescription bottle number in Qualtrics, a HIPAA-compliant online resource that collects, stores, and analyzes data. Demographic information such as age and sex will also be stored in Qualtrics. Each week for one month, patients will be sent an email with a link asking them to complete a Qualtrics survey to report 1) the number of remaining pills, 2) their average pain scale ranging from 1-9, 3) what additional medications they took, if any, and 4) whether they have experienced any medication-related side effects or complications. In this way, we will determine the timing of medication administration for each patient and quantify each patient's level of pain, while assessing for patient safety.

Six months post-injury, patients who sustained tibia fractures will receive repeat X-rays. One final Qualtrics survey will be e-mailed to these patients at this time to determine their average degree of pain on a scale of 1-9, their functional recovery on a scale of 1 to 3 (mild, moderate, or severe impairment) and whether they underwent treatments such as physical therapy or surgery. The survey will also assess for lifestyle factors known to increase nonunion rates including body habitus, medical problems, and other medications taken.

Six months following enrollment, patients who ruptured their Achilles tendon will be sent a link to a Qualtrics survey via email. On this survey, they will be asked 10 questions with responses on a scale of 0 to 10 that comprise the ATRS (29). A higher score (out of 100) indicates better functional outcomes. Patients will also be asked if they underwent treatments such as physical therapy or surgery. Body habitus, medical problems, other medications taken, smoking status, pregnancy status, and fluoroquinolone use will also be assessed on this survey, as these factors may impact tendon recovery.

ELIGIBILITY:
Inclusion:

* Adult patients (over 18) presenting within 24 hours of a tibia fracture
* Adult patients (over 18) presenting within 24 hours of an Achilles tendon rupture

Exclusions:

Patients will be excluded if they:

* have a contraindication to Ibuprofen or Acetaminophen use
* don't have access to e-mail
* require emergent surgery (such as an open fracture)
* have a diagnosis of osteoporosis
* have already taken one of the study drugs since their injury
* are pregnant (due to their inability to take NSAIDs)
* are < 18 years old (due to differences in bone and tendon healing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of non-union after tibia fracture | 6 months
  Fractures
Functional Recovery after Achilles Tendon Rupture | 6 months
  Achilles Tendon Total Rupture Score measures functional recovery after Achilles tendon rupture on a scale of 0 (worse) to 100 (best).

SECONDARY OUTCOMES:
Functional Impairment after Tibia Fracture on a scale of 1 to 3 (none to severe) | 6 months
  The score quantifies functional impairment on a scale of 1 (none) to 3 (severe)
Degree of pain after Tibia Fracture on a scale of 1-9 | 6 months
  The score quantifies pain on a scale of 1 (none) to 9 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Franco, MD PhD, Principal Investigator — Assistant Professor

IPD SHARING:
Plan to Share IPD: No